CLINICAL TRIAL: NCT00138619
Title: Extension to a Study on the Efficacy and Safety of Vildagliptin Compared to Rosiglitazone in Drug Naive Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2327E1
Record Dates: First submitted 2005-08-27; First posted 2005-08-30 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
This is an 80-week extension to a study to assess the safety and effectiveness of vildagliptin, an unapproved drug, compared to rosiglitazone in lowering overall blood glucose levels in people with type 2 diabetes who have not previously been treated with drug therapy to lower their blood sugar. The purpose of the extension study is to gather data on the long-term safety and effectiveness of vildagliptin in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Only patients successfully completing study CLAF237A2327 are eligible
* Written informed consent
* Ability to comply with all study requirements

Exclusion Criteria:

* Premature discontinuation from study CLAF237A2327
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2004-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Safety during 104 weeks of treatment
Change from baseline in HbA1c at 104 weeks

SECONDARY OUTCOMES:
Change in HbA1c between 24 weeks and 104 weeks
Change from baseline in fasting plasma glucose at 104 weeks
Change in fasting plasma glucose between 24 weeks and 104 weeks
Change from baseline in HOMA B at 104 weeks
Change in HOMA B between 24 weeks and 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Investigative Centers, Germany

REFERENCES:
- [Derived] Rosenstock J, Niggli M, Maldonado-Lutomirsky M. Long-term 2-year safety and efficacy of vildagliptin compared with rosiglitazone in drug-naive patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2009 Jun;11(6):571-8. doi: 10.1111/j.1463-1326.2008.01021.x. Epub 2009 Apr 5. PMID 19383032